CLINICAL TRIAL: NCT05291546
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Two-Part, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of REGN9035 (an Anti-REGN5381 Antibody and Reversal Agent) and REGN5381 (an NPR1 Agonist Antibody) When Administered Alone or in Sequence to Healthy Volunteers and Mildly Hypertensive Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of REGN9035 in Healthy Adult Volunteers and Mildly Hypertensive Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R9035-HV-2125; 2021-005174-26 (EudraCT Number)
Record Dates: First submitted 2022-02-28; First posted 2022-03-22 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Mild Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A (Experimental): Single ascending dose (SAD) of REGN9035 or matching placebo given by intravenous (IV) administration.
  Interventions: Drug: REGN9035; Other: Placebo
- Part B (Experimental): Selected doses of REGN5381 or matching placebo given by IV administration followed by selected doses of REGN9035 and/or matching placebo via IV infusion
  Interventions: Drug: REGN9035; Drug: REGN5381; Other: Placebo

INTERVENTIONS:
Drug: REGN9035 — Part A: Single dose administered by IV infusion on day 1. Part B: Selected doses administered by IV infusion on day 2 or 22.
Drug: REGN5381 — Part B: Selected doses administered by IV infusion on day 1.
  Arms: Part B
Other: Placebo — Part A: Single dose administered by IV infusion on day1. Part B: Single dose administered by IV infusion on day 1, day 2 and/or day 22.

SUMMARY:
The primary objective of the study is to:

• Evaluate the safety and tolerability of REGN5381 and REGN9035 administered alone or sequentially.

The secondary objectives of the study are to:

* Evaluate the ability of single intravenous (IV) doses of REGN9035 (compared to placebo) to reverse the acute hemodynamic effects of REGN5381
* Evaluate the hemodynamic effects of single IV doses of REGN5381
* Evaluate the persistence of the hemodynamic effects of single IV doses of REGN5381 and the reversal of REGN5381 effects by REGN9035 (compared to placebo)
* Evaluate the pharmacokinetics of single IV doses of REGN5381 and REGN9035 administered alone or sequentially

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index (BMI) between 18 and 32 kg/m2, inclusive, at the screening visit.
2. Normal or mildly elevated blood pressure as defined in the protocol.

Key Exclusion Criteria:

1. History of unexplained syncope or autonomic dysfunction.
2. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease.
3. Protocol-defined risk factors for cardiovascular disease.

Note: Other protocol defined inclusion / exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment Emergent Adverse Events (TEAEs) | Up to Day 162

SECONDARY OUTCOMES:
Mean systolic blood pressure (SBP) obtained after study drug administration | Up to Day 3
  Up to 24 hours after study drug administration.
Mean diastolic blood pressure (DBP) obtained after study drug administration | Up to Day 3
Mean arterial pressure (MAP) obtained after study drug administration | Up to Day 3
Mean pulse pressure (PP) obtained after study drug administration | Up to Day 3
Mean pulse rate (PR) obtained after study drug administration | Up to Day 3
Mean stroke volume (SV) obtained after study drug administration | Up to Day 3
Absolute change in the mean SBP obtained after study drug administration | Up to Day 3
Absolute change in the mean DBP obtained after study drug administration | Up to Day 3
Absolute change in the mean MAP obtained after study drug administration | Up to Day 3
Absolute change in the mean PP obtained after study drug administration | Up to Day 3
Absolute change in the mean PR obtained after study drug administration | Up to Day 3
Absolute change in the mean SV obtained after study drug administration | Up to Day 3
Maximum change in the mean SBP obtained after study drug administration | Up to Day 3
Maximum change in the mean DBP obtained after study drug administration | Up to Day 3
Maximum change in the mean MAP obtained after study drug administration | Up to Day 3
Maximum change in the mean PP obtained after study drug administration | Up to Day 3
Maximum change in the mean PR obtained after study drug administration | Up to Day 3
Maximum change in the mean SV obtained after study drug administration | Up to Day 3
Percent change in the mean SBP obtained after study drug administration | Up to Day 3
Percent change in the mean DBP obtained after study drug administration | Up to Day 3
Percent change in the mean MAP obtained after study drug administration | Up to Day 3
Percent change in the mean PP obtained after study drug administration | Up to Day 3
Percent change in the mean PR obtained after study drug administration | Up to Day 3
Percent change in the mean SV obtained after study drug administration | Up to Day 3
Absolute change from baseline (post-REGN5381 administration) in the mean SBP obtained after study drug administration | Up to Day 3
Absolute change from baseline (post-REGN5381 administration) in the mean DBP obtained after study drug administration | Up to Day 3
Absolute change from baseline (post-REGN5381 administration) in the mean MAP obtained after study drug administration | Up to Day 3
Absolute change from baseline (post-REGN5381 administration) in the mean PP obtained after study drug administration | Up to Day 3
Absolute change from baseline (post-REGN5381 administration) in the mean PR obtained after study drug administration | Up to Day 3
Absolute change from baseline (post-REGN5381 administration) in the mean SV obtained after study drug administration | Up to Day 3
Maximum change from baseline (post-REGN administration) in the mean SBP obtained after study drug administration | Up to Day 3
Maximum change from baseline (post-REGN administration) in the mean DBP obtained after study drug administration | Up to Day 3
Maximum change from baseline (post-REGN administration) in the mean MAP obtained after study drug administration | Up to Day 3
Maximum change from baseline (post-REGN administration) in the mean PP obtained after study drug administration | Up to Day 3
Maximum change from baseline (post-REN5381 administration) in the mean PR obtained after study drug administration | Up to Day 3
Maximum change from baseline (post-REGN5381 administration) in the mean SV obtained after study drug administration | Up to Day 3
Percent change from baseline (post-REN5381 administration) in the mean SBP obtained after study drug administration | Up to Day 3
Percent change from baseline (post-REN5381 administration) in the mean DBP obtained after study drug administration | Up to Day 3
Percent change from baseline (post-REN5381 administration) in the mean MAP obtained after study drug administration | Up to Day 3
Percent change from baseline (post-REN5381 administration) in the mean PP obtained after study drug administration | Up to Day 3
Percent change from baseline (post-REN5381 administration) in the mean PR obtained after study drug administration | Up to Day 3
Percent change from baseline (post-REN5381 administration) in the mean SV obtained after study drug administration | Up to Day 3
Absolute change from baseline (pre-REGN5381 administration) in the mean SBP obtained after study drug administration | Up to Day 3
Absolute change from baseline (pre-REGN5381 administration) in the mean DBP obtained after study drug administration | Up to Day 3
Absolute change from baseline (pre-REGN5381 administration) in the mean MAP obtained after study drug administration | Up to Day 3
Absolute change from baseline (pre-REGN5381 administration) in the mean PP obtained after study drug administration | Up to Day 3
Absolute change from baseline (pre-REGN5381 administration) in the mean PR obtained after study drug administration | Up to Day 3
Absolute change from baseline (pre-REGN5381 administration) in the mean SV obtained after study drug administration | Up to Day 3
Maximum change from baseline (pre-REGN administration) in the mean SBP obtained after study drug administration | Up to Day 3
Maximum change from baseline (pre-REGN administration) in the mean DBP obtained after study drug administration | Up to Day 3
Maximum change from baseline (pre-REGN administration) in the mean MAP obtained after study drug administration | Up to Day 3
Maximum change from baseline (pre-REGN administration) in the mean PP obtained after study drug administration | Up to Day 3
Maximum change from baseline (pre-REGN administration) in the mean PR obtained after study drug administration | Up to Day 3
Maximum change from baseline (pre-REGN administration) in the mean SV obtained after study drug administration | Up to Day 3
Percent change from baseline (pre-REN5381 administration) in the mean SBP obtained after study drug administration | Up to Day 3
Percent change from baseline (pre-REN5381 administration) in the mean DBP obtained after study drug administration | Up to Day 3
Percent change from baseline (pre-REN5381 administration) in the mean MAP obtained after study drug administration | Up to Day 3
Percent change from baseline (pre-REN5381 administration) in the mean PP obtained after study drug administration | Up to Day 3
Percent change from baseline (pre-REN5381 administration) in the mean PR obtained after study drug administration | Up to Day 3
Percent change from baseline (pre-REN5381 administration) in the mean SV obtained after study drug administration | Up to Day 3
Percentage of participants who return to within 10% of baseline (pre-REGN5381 administration) SBP obtained after study drug administration. | Baseline to Day 3
Percentage of participants who return to within 10% of baseline (pre-REGN5381 administration) DBP obtained after study drug administration. | Baseline to Day 3
Percentage of participants who return to within 10% of baseline (pre-REGN5381 administration) MAP obtained after study drug administration. | Baseline to Day 3
Percentage of participants who return to within 10% of baseline (pre-REGN5381 administration) PP obtained after study drug administration. | Baseline to Day 3
Percentage of participants who return to within 10% of baseline (pre-REGN5381 administration) PR obtained after study drug administration. | Baseline to Day 3
Percentage of participants who return to within 10% of baseline (pre-REGN5381 administration) SV obtained after study drug administration. | Baseline to Day 3
Time to return to within 10% of baseline (pre-REGN5381) SBP | Up to approximately Day 162
Time to return to within 10% of baseline (pre-REGN5381) DBP | Up to approximately Day 162
Time to return to within 10% of baseline (pre-REGN5381) MAP | Up to approximately Day 162
Time to return to within 10% of baseline (pre-REGN5381) PP | Up to approximately Day 162
Time to return to within 10% of baseline (pre-REGN5381) PR | Up to approximately Day 162
Time to return to within 10% of baseline (pre-REGN5381) SV | Up to approximately Day 162
SBP | Through Day 36
DBP | Through Day 36
MAP | Through Day 36
PP | Through Day 36
PR | Through Day 36
Absolute change from baseline in SBP | Through Day 36
Absolute change from baseline in DBP | Through Day 36
Absolute change from baseline in MAP | Through Day 36
Absolute change from baseline in PP | Through Day 36
Absolute change from baseline in PR | Through Day 36
Percent change from baseline in SBP | Through Day 36
Percent change from baseline in DBP | Through Day 36
Percent change from baseline in MAP | Through Day 36
Percent change from baseline in PP | Through Day 36
Percent change from baseline in PR | Through Day 36
Concentrations of total REGN9035 | Up to Day 162
Concentrations of total REGN5381 over time | Up to Day 162
Concentrations of total REGN9035 and/or total REGN5381 | Up to Day 162

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- Universitair Ziekenhuis Leuven Gasthuisberg Campus, Leuven, Belgium
- Charite Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org